CLINICAL TRIAL: NCT06693778
Title: Utilizing Electronic Clinical Decision Support to Enhance mTBI Care at the Primary Care Point of Entry
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 22-020695; U01CE003479 (NIH)
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury
Keywords: Clinical Decision Support; Persisting Post-Concussion Symptoms
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Select Primary Care Practices: Select pediatric primary care practices (3 urban and 3 suburban) that are evaluating patients for mild traumatic brain injury with an electronic clinical decision support tool.
  Interventions: Other: electronic Clinical Decision Support tool for risk stratification of pediatric patients with mTBI
- Comparison Primary Care Practices: Pediatric primary care practices that are NOT using the electronic clinical decision support tool to evaluate patients for mild traumatic brain injury.

INTERVENTIONS:
Other: electronic Clinical Decision Support tool for risk stratification of pediatric patients with mTBI — eCDS tool for risk stratification of pediatric mTBI patients
  Groups: Select Primary Care Practices

SUMMARY:
Six primary care practices within a large Philadelphia pediatric care network will use an electronic Clinical Decision Support (eCDS) tool as standard care for concussion evaluation. The eCDS tool will include a prediction rule for children aged 5-18 assessed for mild traumatic brain injury (mTBI). The eCDS tool predicts risk for persistent symptoms and prompts referral to specialty care for those deemed high risk. This research proposes to analyze the clinical and process outcomes in these six practices relative to the rest of the care network, specifically, whether the eCDS tool reduces time to symptom resolution.

DETAILED DESCRIPTION:
The electronic Clinical Decision Support tool will include a prediction rule for children aged 5-18 assessed for mild traumatic brain injury (mTBI). It predicts risk for persistent symptoms and prompts referral to specialty care for those who are high-risk. The eCDS tool consists of a validated, age-appropriate symptom scale, risk stratification with indication for specialty referral, personalized return to activity guidance based on symptom exacerbation, and guidance on minimizing prolonged rest and promoting active management.

Each year for three years, the eCDS tool will go live at a new pair of sites (1 urban, 1 suburban). Training will be provided to the primary care providers at these sites on utilizing the eCDS tool. Anonymous questionnaires will be administered among providers who used the eCDS tool in order to evaluate its appropriateness and acceptability. Interviews will be conducted with a subset of providers to obtain more detailed feedback on the eCDS tool. A medical record review will be conducted of mTBI patients evaluated with the eCDS tool.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 year old patients evaluated for mild Traumatic Brain Injury at a Children's Hospital of Philadelphia primary care practice within the study timeframe

Exclusion Criteria:

* Evidence of moderate or severe TBI

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Head injury patients seen at select primary care practices within the Children's Hospital of Philadelphia network during the study timeframe.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Days until return to symptom baseline | Up to 1 year post-injury
  Review of medical records to determine when patient is considered clinically recovered (number of days to return to pre-injury level of symptoms)

SECONDARY OUTCOMES:
Provider-defined appropriateness of the electronic Clinical Decision Support (eCDS) risk stratification tool | Approximately one year after the eCDS tool is implemented at a primary care location
  Mean System Usability Score (SUS) out of 100 with greater than or equal to 70 defined as acceptable appropriateness. The SUS questionnaire is administered through REDCap and consists of 5 negatively worded statements and 5 positively worded statements about the eCDS tool. Response options range from 1 (Strongly Disagree) to 5 (Strongly Agree). Standard SUS scoring is used to calculate a mean score: negatively worded items are scored as scale value minus 1; positively worded items are scored as 5 minus the scale value. The 10 items are summed and then multiplied by 2.5.
Provider-defined acceptability of the electronic Clinical Decision Support (eCDS) risk stratification tool | Approximately one year after the eCDS tool is implemented at a primary care location
  Providers will complete a questionnaire evaluating the acceptability of the eCDS tool. This questionnaire consists of 10 statements derived from the Technology Acceptance Model with response options ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
Incidence of Persisting Post-Concussion Symptoms (PPCS) | 28 days post-injury
  Number of participants experiencing persistence of at least 3 concussion symptoms above the pre-injury state, 28 days or more post-injury as determined by chart review.
Provider fidelity to the electronic Clinical Decision Support (eCDS) tool | 28 days post-injury
  Percent of patients for whom the provider followed the eCDS tool recommendation. Of the total number of patients the eCDS tool classifies as high risk, how many receive referrals to specialty care (provider fidelity) and how many do not (provider non-fidelity)? Of the total number of patients the eCDS tool classifies as low risk, how many do not receive referrals to specialty care (provider fidelity) and how many do receive referrals (provider non-fidelity)?
Patient adherence to provider recommendations | 3 months post-injury
  Of all patients who received a referral to specialty care, how many scheduled and attended a specialty care appointment, defined as at least 1 interaction with a specialty provider either in person or via telehealth during the acute study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristy Arbogast, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Root JM, Gai J, Sady MD, Vaughan CG, Madati PJ. Identifying Risks for Persistent Postconcussive Symptoms in a Pediatric Emergency Department: An Examination of a Clinical Risk Score. Arch Clin Neuropsychol. 2022 Jan 17;37(1):30-39. doi: 10.1093/arclin/acab032. PMID 33993203
- [Background] Sutton RT, Pincock D, Baumgart DC, Sadowski DC, Fedorak RN, Kroeker KI. An overview of clinical decision support systems: benefits, risks, and strategies for success. NPJ Digit Med. 2020 Feb 6;3:17. doi: 10.1038/s41746-020-0221-y. eCollection 2020. PMID 32047862